CLINICAL TRIAL: NCT04178083
Title: Comparison of Postoperative Results of Laparoscopic Sacrohysteropexy, Modified Laparoscopic Lateral Suspension and Laparoscopic Pectopexy in Patients With Uterine Prolapse.
Brief Title: Comparison of Laparoscopic Sacrohysteropexy, Modified Laparoscopic Lateral Suspension and Laparoscopic Pectopexy.
Status: Completed | Type: Observational
Sponsor: Diyarbakir Women's and Children's Diseases Hospital (Other)
Responsible Party: Principal Investigator, Şerif AKSİN, Medical Doctor, Diyarbakir Women's and Children's Diseases Hospital
Other Study IDs: DiyarbakirWCDH 2
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Pelvic Organ Prolapse; Laparoscopy
Keywords: laparoscopy; pelvic organ prolapse; modified lateral süspension; pectopexy; sacrohysteropexy; hysteropexy; sacropexy; cervicopexy; sacrocervicopexy
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laparoscopic Sacrohysteropexy,: Under general anesthesia,laparoscopic approach is used to enter the abdomen.Following this, visceral peritoneum is held with forceps from the point where the sacro-uterine ligaments adhere to the uterus.
  cut with unipolar scissors to the sacrouterin ligaments approximately 2-4 cm in the midline a transverse incision is made and the posterior wall of the cervix is reached. Approx. 10-15 x2 cm polypropylene mesh 5 mm trocar is inserted into the abdomen with the help of grasper and one end three points with 2/0 non-absorbable prolene sutures in the midline cervix Intracorporeal suture technique.
  After the sacral promontorium on peritona about 2 The transverse incision is made to the normal anatomical position and the appropriate mesh length is determined and the other end is fixed to the area prepared on the sacral promontorium at 3 points with 2-0 prolene. Bleeding reperitonization according to intracorporeal suture technique with 2/0 vicry
  Interventions: Diagnostic Test: medical examination
- Modified Laparoscopic Lateral Suspension: A 10 cm diameter trocar is passed through a 1 cm infraumbical incision. In addition, two 5 mm diameter trocar are placed on 4 cm on both sides of the spinal iliac crest, and a 5 mm diameter trocar is placed laterally in the rectus muscle at the left lateral level of the umbilicus. A Prolene network of 25 cm in length is prepared. Dissection of the uterine cavity is performed to expose a mustache. The bottom of the web is secured by suturing the web in the midline and sides of the web with 2-0 prolene. The left and right modified lateral ports are then removed by moving under the bottom of the planet with the help of the planet until the isthmus reaches the bottom of the round ligament. The lateral ports are again slid onto the mesh, placed and sutured with peritoneal 2-0 vicryil, the mesh ends are cut at the skin level and the procedure is terminated.
  Interventions: Diagnostic Test: medical examination
- Laparoscopic Pectopexy: First, the peritoneal layer on the top and side of the bladder opens parallel to the round ligament toward the right pelvic sidewall.
  The iliopectineal ligament is then located under the guidance of the obliterated umbilical artery, lateral to the obliterated umbilical artery and medially of the outer iliac vein.
  iliopectineal (Cooper) ligament exposing a segment of approximately 3-4 cm is formed.
  After completion of the dissections, the ends of the mesh are sutured to both iliopectineal ligaments by intracorporeal suture using nonabsorbable sutures. The middle of the net is fixed with three sutures to the lower anterior segment of the uterus. The peritoneum on the mesh is sutured with an absorbable suture material.
  Interventions: Diagnostic Test: medical examination

INTERVENTIONS:
Diagnostic Test: medical examination — medical examination
  Other Names: Routine gynecological examination for POP-Q

SUMMARY:
The aim of this study was to compare the results of laparoscopic sacrohysteropexy, laparoscopic modified lateral suspens9ion and laparoscopic pectopexy between January 2017 and December 2019 in our clinic.(Patients with at least 12 months of the date of surgery will be called for examination.)

DETAILED DESCRIPTION:
The aim of this study was to compare the results of laparoscopic sacrohysteropexy, laparoscopic modified lateral suspens9ion and laparoscopic pectopexy between January 2017 and December 2019 in our clinic.(Patients with at least 12 months of the date of surgery will be called for examination.)

We will evaluate Pelvic Organ Prolapse Quantitative System (POP-Q), Prolapse Quality of Life Questionnaire (PQoL), Pelvic Organ Prolapse Symptom Score (POP-SS), Visual Analogue Score (VAS), routine gynecologic USG, failure, complication, operation time .

ELIGIBILITY:
Inclusion Criteria:

* patients requiring surgical treatment for the symptomatic stage of pelvic organ prolapse ≥ 2

Exclusion Criteria:

* Age > 70 years
* Severe cardiovascular or respiratory disease
* Pregnancy

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: patients who underwent surgical prolapse uteri operation in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Anatomical improvement according to POP-Q score | 12 months after intervention
  a system for assessing the degree of prolapse of pelvic organs

SECONDARY OUTCOMES:
Change from baseline Prolapse Quality of Life questionnaire (PQoL) to measure quality of life according to pelvic organ prolapse | 12 months after intervention
  The survey includes 20 questions grouped in chapters (areas) related to a specific aspect of quality of life
Change from baseline Pelvic Organ Prolapse Symptom Score (POP-SS) to measure quality of life according to pelvic organ prolapse | 12 months after intervention
  measures the effect of changes in pelvic organ prolapse on quality of life
Change from baseline Visual Analog Score (VAS) for pain | 12 months after intervention
  Participant describes the pain related to the mesh
Failure (%) | 12 months after intervention
  Recurrence rate
Complications | 12 months after intervention
  İnjury

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Principal Investigator — Yes
Locations (1):
- Diyarbakır Women's and Children's Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Veit-Rubin N, Dubuisson JB, Gayet-Ageron A, Lange S, Eperon I, Dubuisson J. Patient satisfaction after laparoscopic lateral suspension with mesh for pelvic organ prolapse: outcome report of a continuous series of 417 patients. Int Urogynecol J. 2017 Nov;28(11):1685-1693. doi: 10.1007/s00192-017-3327-2. Epub 2017 Apr 17. PMID 28417156
- [Background] Bojahr B, Tchartchian G, Waldschmidt M, Ohlinger R, De Wilde RL. Laparoscopic sacropexy: a retrospective analysis of the subjective outcome in 310 cases. Obstet Gynecol Int. 2012;2012:538426. doi: 10.1155/2012/538426. Epub 2011 Sep 7. PMID 21912552
- [Background] Noe KG, Schiermeier S, Alkatout I, Anapolski M. Laparoscopic pectopexy: a prospective, randomized, comparative clinical trial of standard laparoscopic sacral colpocervicopexy with the new laparoscopic pectopexy-postoperative results and intermediate-term follow-up in a pilot study. J Endourol. 2015 Feb;29(2):210-5. doi: 10.1089/end.2014.0413. Epub 2014 Nov 20. PMID 25350228